CLINICAL TRIAL: NCT01940250
Title: A Randomized, Placebo-controlled, Double-blind Trial of Intravenous Magnesium Sulfate for the Management of Severe Hand, Foot and Mouth Disease With Autonomic Nervous System Dysregulation in Vietnamese Children.
Brief Title: Magnesium Sulphate for Severe Hand, Foot and Mouth Disease in Vietnam
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Oxford University Clinical Research Unit, Vietnam (Other)
Collaborators: Hospital for Tropical Diseases, Ho Chi Minh City, Vietnam (Other); Children's Hospital Number 1, Ho Chi Minh City, Vietnam (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 02EI
Record Dates: First submitted 2013-08-22; First posted 2013-09-12 (Estimated); Last update posted 2017-03-07 (Actual); Status verified 2014-11

CONDITIONS: Hand, Foot and Mouth Disease
Keywords: Hand, foot and mouth disease; Autonomic nervous system dysregulation; Magnesium sulphate
MeSH Terms: conditions — Hand, Foot and Mouth Disease | interventions — Magnesium Sulfate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sterile water (Placebo Comparator): Sterile water will be packaged identically to the active comparator.
  Each patient randomized to the placebo arm of the trial will receive a loading dose of 0.5ml/kg intravenous over 20 minutes , followed by a maintenance dose of 0.3 ml/kg/hr to 0.5 ml/kg/hr randomly adjusted by an independent doctor to mimic adjustments made in the active comparator arm for 72 hrs.
  Interventions: Drug: Sterile water
- Magnesium sulphate (Active Comparator): Each patient randomized to the treatment arm of the trial will receive a loading dose of 50mg/kg intravenous over 20 minutes (0.5ml/kg), followed by a maintenance dose of 30-50 mg/kg/hr (0.3 ml/kg/hr to 0.5 ml/kg/hr) for 72 hrs.
  The maintenance dose will be determined by increasing the loading infusion dose 0.1 ml/kg/hr (10mg/kg/hr) every 15 minutes to a maximum dose of 0.5 ml/kg/hr (50 mg/kg/hr), with the following caveats:
  * If the systolic BP decreases to < 90th percentile for age, gender and length the dose will be reduced by 1 stage every 15 mins
  * If the systolic BP increases to the levels detailed in the study protocol for treatment failure, action will be taken as indicated
  * If the systolic BP decrease rapidly more than 25% over 15 minutes
  * If the plasma Mg level > 2.5 mmol/l or < 1.8 mmol/l a 25% increase or decrease in the infusion rate will be implemented as appropriate.
  Interventions: Drug: Magnesium Sulphate

INTERVENTIONS:
Drug: Magnesium Sulphate — MgSO4 IV infusion
  Other Names: magnesi sulfat krabi 15%
  Arms: Magnesium sulphate
Drug: Sterile water — H2O IV infusion
  Arms: Sterile water

SUMMARY:
Hand foot and mouth disease (HFMD) is a common infectious disease caused by a number of different viruses - a small proportion of children infected with a particular type of enterovirus (EV71) develop neurological and systemic complications that may prove fatal. Very large epidemics of EV71 related HFMD have occurred across Asia in recent years; in 2011, in excess of 100,000 Vietnamese children were diagnosed with HFMD and 164 died.

In children with severe HFMD the particular part of the brain that regulates the heart, blood circulation, and breathing responses can be affected. Management of this complication is very difficult and we currently use an expensive drug (milrinone) that is hard to obtain and has significant side effects, without having good evidence that it is effective.

Magnesium sulphate (Mg) is a cheap, readily available drug that has been used in other diseases with similar complications, and we have preliminary data from a small case series that suggests it might be a good treatment for HFMD patients with signs indicating this type of brain involvement.

We think that early intervention with Mg, when signs of brain involvement are still relatively mild, will control this problem better than waiting until it is well established and giving milrinone as at present, and this in turn may prevent progression to severe disease. The aims of the project are to evaluate the effects of Mg on hypertension, signs of brain dysfunction, outcome (death or neurological sequelae), changes in a variety of blood and urine components, and measures of cardiovascular function, in severe HFMD.

The study design is a randomized double-blind placebo-controlled clinical trial. Children on the pediatric intensive care unit with a clinical diagnosis of hand, foot and mouth disease will be eligible for enrolment if the blood pressure exceeds the internationally recognized threshold for Stage 1 hypertension, they exhibit at least one other sign of brain stem dysfunction, and there is written informed consent by a parent or guardian.

According to the randomization, patients will receive an initial loading dose followed by a maintenance infusion, of either Mg or identical placebo for 72 hours; all staff involved in patient care will remain unaware of the treatment allocation, but staff from another department will monitor Mg blood levels to ensure safety and adequate dosing. A total of 190 patients (95 in each arm) will be recruited.

DETAILED DESCRIPTION:
Background:

Hand foot and mouth disease (HFMD) is a common infectious disease caused by a variety of enteroviruses. A small proportion of those infected with enterovirus 71 (EV71) develop neurological and systemic complications that may prove fatal. Over the past 15 years EV71 related HFMD has caused increasing epidemics of HFMD across Asia; in 2011, in excess of 100,000 Vietnamese children were diagnosed clinically with HFMD and 164 died. The neurological problem of most concern is brainstem encephalitis, causing autonomic nervous system (ANS) dysregulation that may progress rapidly to cardiopulmonary failure. Management of ANS dysregulation is difficult even in sophisticated western intensive care units. The phosphodiesterase-3 inhibitor, Milrinone, was reported to control hypertension and support myocardial function in a small informal study of severe HFMD compared to historical controls, but in practice treatment remains largely empirical. ANS dysregulation also occurs in severe tetanus and there is a body of evidence indicating that intravenous magnesium sulphate (Mg) is effective in controlling tetanus-associated cardiovascular instability. Mg is also used widely for eclampsia, severe asthma and pulmonary hypertension, and there are reports of rapid control of life-threatening autonomic hyperreflexia in patients with spinal lesions. Formal safety data in children are limited, but adverse effects appear to be infrequent. In a series of 24 severe EV71 confirmed HFMD cases managed recently at the Hospital for Tropical Diseases, Ho Chi Minh City, Mg was added when hypertension remained poorly controlled despite high-dose Milrinone. In all cases the blood pressure (BP) reduced within 30-60 minutes and remained stable subsequently on a continuous Mg infusion for 48-72 hours.

Hypothesis and Aims:

We hypothesize that early intervention with Mg, when ANS dysregulation first becomes apparent, will control cardiovascular instability and prevent progression to severe disease. The main aims are as follows:-

* To evaluate the effects of Mg on hypertension and ANS dysregulation in severe HFMD
* To evaluate the effects of Mg on outcome (death or neurological sequelae) in severe HFMD
* To evaluate changes in plasma/urine catecholamine levels, cardiac output and systemic vascular resistance (SRV) in severe HFMD, and to assess the impact of Mg on these parameters.

Study Design:

We plan a randomized double blind trial comparing intravenous Mg with placebo in children admitted to the pediatric intensive care unit with clinical HFMD, ANS dysregulation, and Stage 1 hypertension. Patients will be eligible for enrolment if the arterial blood pressure exceeds the 95th centile for age, gender and length/height for at least 30 minutes while the child is not distressed, they exhibit at least one other criterion for ANS dysregulation, and a parent/guardian gives written informed consent. Specific renal and cardio-respiratory exclusion criteria will apply.

A loading dose of 50mg/kg of either Mg or identical placebo will be given over 20 minutes followed by a maintenance infusion for 72 hours according to response, aiming for Mg levels 2-3 times normal in the treatment arm. All staff involved in clinical care will be blind to the treatment allocation, and Mg levels will be monitored and adjusted by independent doctors from another clinical facility.

The primary endpoint will be a composite endpoint of disease progression defined as occurrence of any of the following within 72 hours: specific blood pressure criteria necessitating addition of milrinone, need for ventilation, development of shock, or death. Secondary endpoints will include presence of neurological sequelae at discharge in survivors, and various measures of cardiac output and systemic vascular resistance, catecholamine and cytokine levels.

Based on 1:1 randomization, an anticipated relative reduction of the risk of progression of 50% (from 50% in the control arm to 25% in Mg recipients, information from our case series plus indirect evidence from studies on severe tetanus), 90% power and a two-sided 5% significance level, 85 patients per treatment group are required. To allow for some violations of our assumptions and losses to follow-up, we plan to recruit 190 patients (95 patients per treatment arm) into the study.

Potential Impact:

Given the very large numbers of HFMD cases being seen in hospitals in Asia currently, if Mg is shown to be effective in controlling ANS dysregulation and preventing severe HFMD complications this would be of major importance for paediatric care throughout the Asian region. Mg is cheap, readily available and safe whereas milrinone is expensive, has a significant side effect profile and is often not available outside major centres.

ELIGIBILITY:
Inclusion Criteria:

* Age 6 months to 15 years
* Clinical suspicion of HFMD requiring PICU/HDU admission
* Considered severe enough to warrant invasive blood pressure monitoring by PICU/HDU staff
* Development of hypertension defined as follows:

  * For children aged 1 year and over, at least 3 consecutive systolic blood pressure recordings above the 95th centile for age, gender and length (USA guidelines for defining Stage 1 hypertension in children, (Appendix 2)) measured invasively over a period of 20 minutes provided the child is not distressed or crying [30, 31].
  * For children aged 6 months to 1 year, systolic BP > 100 mm Hg measured invasively on at least 3 occasions over a period for 20 minutes provided the child is not distressed or crying
* Plus one or more of the following criteria:

  * Tachypnoea for age
  * Irregular or labored breathing, but with SpO2 above 92% in air and normal ABG (pH, pCO2, pO2, HCO3 all within the normal range for the local laboratory)
  * Resting heart rate > 150 bpm
  * Mottled skin
  * Profuse sweating
  * Refractory fever
  * Hyperglycemia
* Informed consent

Exclusion Criteria:

* Past history of hypertension, chronic renal, cardiac or pulmonary disease, or any neurological disorder
* Hypertensive emergency
* Already commenced milrinone or any other inotropic agents
* Respiratory distress with SpO2<92% in air or PaCO2>45 mm Hg
* AV block or any arrhythmia
* Acute renal failure

Ages: 6 Months to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 26 (Actual)
Dates: Start 2014-04-21 (Actual); Primary Completion 2016-06-30 (Actual); Study Completion 2016-12-28 (Actual)

PRIMARY OUTCOMES:
Number of patients who experience at least one of the clinical events listed below (composite endpoint) | 72 hours after start of study drug infusion
  Number of patients who meet one or more of the following criteria:
  1. Blood pressure criteria necessitating addition of milrinone following Vietnam Ministry of Health guidelines for the treatment of hand, foot and mouth disease
  2. Need for mechanical ventilation
  3. Development of shock
  4. Death

SECONDARY OUTCOMES:
Death | 72 hours after start of study drug infusion
Blood pressure criteria necessitating addition of milrinone following Vietnam Ministry of Health guidelines for the treatment of hand, foot and mouth disease | 72 hours after start of study drug infusion
Need for mechanical ventilation | 72 hours after start of study drug infusion
  According to Viet Nam Ministry of Health guidelines: Ventilation Criteria:
  If a patient continues to display any of the following criteria despite oxygenation via nasal cannula and cardiac support with inotropic drugs for more than 60 minutes.
  * Labored breathing
  * Tachypnea with resting respiratory rate > 70 / minute without fever
  * Hypoxemia and/or fluctuating SpO2
  * Poor tissue perfusion and persistent resting heart rate > 180 beats/minute without fever
  Or
  * Decorticate or decerebrate rigidity
  * Coma (Glasgow Coma Scale < 10 )
Development of shock | 72 hours after start of study drug infusion
Requirement for inotropic agents (eg dobutamine) | During hospital admission - expected average length of admission 5 days
  If heart rate> 170 beats/minute
Presence of neurological sequelae at discharge in survivors | At hospital discharge - expected average discharge day 5
  Number of surviving patients who have neurological sequelae at hospital discharge
Neurodevelopmental status | 6 months
  Measured by . Children 36 months and under at enrollment will use the Bayley infant scales of development III. Children 48 months and above at enrollment will use the Movement ABC-2 tool for their assessments. The children aged between 37 and 47 months at enrolment will have both assessments done at both visits.
Duration of hospitalization | At hospital discharge - expected average discharge day 5
  Number of days from study enrollment to discharge
Number of adverse events and serious adverse events | During hospital admission - expected average length of admission 5 days
  Number of adverse events and severe adverse events that occur in the two treatment arms during hospitalization.

CONTACTS AND LOCATIONS:
Overall Officials: Bridget Wills, MD, Principal Investigator — Oxford University Clinical Research Unit
Locations (2):
- Vietnam (2):
  - Children's Hospital 1, Ho Chi Minh City
  - Hospital for Tropical Diseases, Ho Chi Minh City

REFERENCES:
- [Derived] Phan QT, Phung LK, Truong KH, Huynh TT, Pham GT, Nguyen BN, Tran QT, Huynh VNT, Nguyen TTM, Le TPK, Le NNT, Sabanathan S, van Doorn HR, Van Le T, Nguyen TD, Merson L, Nguyen DTP, Geskus R, Nguyen HT, Nguyen CVV, Wills B. Assessing the efficacy and safety of magnesium sulfate for management of autonomic nervous system dysregulation in Vietnamese children with severe hand foot and mouth disease. BMC Infect Dis. 2019 Aug 22;19(1):737. doi: 10.1186/s12879-019-4356-x. PMID 31438878
- [Derived] Qui PT, Khanh TH, Trieu HT, Giang PT, Bich NN, Thoa le PK, Nhan le NT, Sabanathan S, Van Doorn R, Toan ND, Merson L, Dung NT, Khanh LP, Wolbers M, Hung NT, Chau NV, Wills B. Intravenous magnesium sulfate for the management of severe hand, foot, and mouth disease with autonomic nervous system dysregulation in Vietnamese children: study protocol for a randomized controlled trial. Trials. 2016 Feb 19;17:98. doi: 10.1186/s13063-016-1215-6. PMID 26896318
- See also: Oxford University Clinical Research Unit, Viet Nam — http://www.oucru.org